CLINICAL TRIAL: NCT04807478
Title: A Multicenter, Prospective, Controlled, Longitudinal-Cohort Study Assessing the Safety of Omegaven in Pediatric Patients With Parenteral Nutrition-Associated Cholestasis (PNAC)
Brief Title: Safety of Omegaven in Pediatric Patients With Parenteral Nutrition-Associated Cholestasis (PNAC)
Status: Withdrawn | Type: Observational
Why Stopped: New study protocol under development
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: OMEG-038-CP4
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Parenteral Nutrition Associated Liver Disease; Essential Fatty Acid Deficiency; Neurocognitive Deficit; Malnutrition; Pediatric ALL
MeSH Terms: conditions — Malnutrition; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fish oil triglycerides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients: Pediatric patients with new-onset PNAC
  Interventions: Drug: Omegaven® (fish oil triglycerides) Injectable Emulsion

INTERVENTIONS:
Drug: Omegaven® (fish oil triglycerides) Injectable Emulsion — Dose, frequency and duration is a decision of the Investigator

SUMMARY:
This study will demonstrate Short-, mid-, and long-term safety in pediatric patients with Parenteral Nutrition-Associated Cholestasis treated with Omegaven®, which is indicated as a source of calories and fatty acids in this patient population

DETAILED DESCRIPTION:
Prospective, controlled, longitudinal-cohort phase IV study to assess safety of Omegaven in Pediatric Patients with PNAC, in order to demonstrate short-, mid-, and long-term safety with respect to EFAD, serious bleeding events, life-threatening pleural and pericardial effusions, and neurocognitive development. Pediatric patients with PNAC receiving Omegaven as part of their routine nutritional management will be compared to those treated with another FDA-approved ILE for pediatric patients. Patients who are switched to a non-FDA-approved ILE or to Omegaven will be analyzed separately. Use of ILE will be as indicated by their treating physician, ideally for ≥ 1 year. Dosing modalities are to be taken from the pertinent prescribing information.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent(s) or legal guardian(s) has provided a signed and dated Informed Consent Form (ICF).
2. Patient is PN-dependent and within the past 21 days has been diagnosed with PNAC, defined as direct or conjugated bilirubin (DBil) ≥ 2.0 mg/dL with no other known cause of liver dysfunction at the time of enrollment.
3. Patient has feeding intolerance or at least one gastrointestinal disorder requiring PN.
4. Patient is < 6 months corrected age (expected time of delivery to time of screening).

Exclusion Criteria:

1. Patient has any other known cause of chronic liver disease such as hepatitis C, cystic fibrosis, biliary atresia, alpha-1-antitrypsin deficiency, passive hepatic congestion due to heart failure, etc.
2. Patient has known cirrhosis (liver biopsy is not required under this protocol).
3. Patient has known portal vein thrombosis (imaging studies are not required under this protocol).
4. Patient has previously received a liver-only or liver-inclusive transplant.
5. Patient has a major cardiac anomaly with hemodynamic instability.
6. Patient has a major life-threatening disease (e.g., sepsis requiring high-dose vasopressors, acute respiratory distress syndrome, veno-occlusive disease, cancer).
7. Patient has multi-organ failure, septic shock, hypotension requiring pressor therapy, persistent pulmonary hypertension requiring inhaled nitric oxides, or requires extracorporeal membrane oxygenation (ECMO) or similar intervention.
8. Patient has renal failure and requires dialysis.
9. Patient has a severe hemorrhagic disorder.
10. Patient has an INR > 2.0.
11. Patient has severe hyperlipidemia or a severe disorder of lipid metabolism characterized by hypertriglyceridemia (i.e., serum triglyceride level > 1,000 mg/dL).
12. Patient has a record of a previous T:T ratio ≥ 0.2 or had a previous diagnosis of EFAD.
13. Patient has a central nervous system anomaly (e.g., anencephaly) or any injury (e.g., grade 3 or 4 intraventricular hemorrhage, moderate to severe hypoxic ischemic encephalopathy) that will affect neurodevelopment.
14. Patient has been diagnosed with or is suspected to have a genetic disorder known to be associated with neurodevelopmental impairment (e.g., trisomy 21, 18, 13).
15. Patient has been diagnosed with or is suspected to have an inborn error of metabolism.
16. Patient has a known hypersensitivity to fish or egg protein or to any of the active ingredients or excipients of Omegaven.
17. Patient's medical care has been deemed futile by the medical team.
18. Patient is enrolled in any other study with an investigational medicinal product.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female pediatric patients < 6 months old (corrected age) with new-onset PNAC (diagnosed within the past 21 days) will be enrolled at multiple sites; PNAC is defined as being PN-dependent with a DBil level ≥ 2.0 mg/dL and no other known cause of liver dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of: | Through study completion, a maximum of 6 years
  1. Incidence of EFAD
  2. Incidence of serious bleeding events
  3. Incidence of life-threatening pericardial effusion events
  4. Incidence of life-threatening pleural effusion events
  5. Severity of any neurodevelopmental delays.

OTHER OUTCOMES:
Adverse events (AEs)/serious adverse events (SAEs) | Through study completion, a maximum of 6 years
  The incidence of adverse events (AEs)/serious adverse events (SAEs)